CLINICAL TRIAL: NCT07082049
Title: A Randomized Controlled Trial on Artificial Intelligence-Powered Large Language Model-Assisted Doctor-Patient Preoperative Communication for Psychological Distress Alleviation and Healthcare Efficiency Improvement in Prostate Cancer Patients
Brief Title: AI-LLM Communication Aid in Prostate Cancer Care (AI-CAP）
Acronym: AI-CAP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Bo Dai, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FUSCC-AI-CAP
Record Dates: First submitted 2025-06-10; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; large language model; anxiety; patient distress; healthcare efficiency
MeSH Terms: conditions — Prostatic Neoplasms; Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLM-assisted (Experimental): Patients will communicate with the LLM before surgery, which will provide answers based on their various concerns, including diagnosis, surgical plan selection, surgery risks, and handling of complications. Subsequently, patients will also continue to participate in the routine pre-operative communication held by surgeons.
  Interventions: Procedure: Prostate surgery; Behavioral: LLM-assisted communication; Behavioral: Routine preoperative communication
- Conventional routine communication (Experimental): Patients will participate routine pre-operative communication, held by the surgical team's lead physician, to inform the patient about the surgical plan selection, surgery risks, and the situation regarding post-operative complications, as well as to answer any patient inquiries.
  Interventions: Procedure: Prostate surgery; Behavioral: Routine preoperative communication

INTERVENTIONS:
Procedure: Prostate surgery — Including but not limited to open radical prostatectomy, laparoscopic radical prostatectomy (LapRP) and robot-assisted radical prostatectomy (RARP).
Behavioral: LLM-assisted communication — Preoperatively, patients will communicate with the LLM, which will provide direct answers to their various questions, including but not limited to diagnosis, treatment options, operative risks, and complication management. To ensure the accuracy of LLM-generated responses in real-world clinical settings, all answers will undergo verification by the researchers before being provided to patients.
  Arms: LLM-assisted
Behavioral: Routine preoperative communication — Preoperatively, patients will attend a consultation with the attending surgeon and surgical team. This physician-led communication will comprehensively discuss, current disease status, treatment options, operative risks, potential complication. The surgical team will subsequently address patient inquiries, followed by executing the informed consent form.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of large language model (LLM)-assisted communication on psychological distress alleviation and healthcare efficiency improvement in prostate cancer patients. The main questions it aims to answer are:

Does LLM-assisted communication reduce preoperative anxiety and negative emotion more effectively than standard care? Can LLM-assisted communication decrease clinician workload while maintaining communication quality?

Researchers will compare the intervention group (LLM-assisted communication) with the control group (standard communication) to see:

Whether LLM-assisted communication has greater reductions in patients' emotional distress scales and physiological stress metrics.

How it impacts clinician workload and communication time.

Participants will:

Undergo baseline assessments before communication, including a range of emotional scales and physiological metrics.

Receive clinician-reviewed LLM-generated materials and/or standard communication before surgery.

Complete assessments after preoperative communication.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed prostate adenocarcinoma confirmed by histopathology;
2. Age 18 years or older;
3. Must be a candidate for radical prostatectomy, including but not limited to laparoscopic radical prostatectomy (LapRP) and robot-assisted radical prostatectomy (RARP);
4. Ability to independently complete questionnaire filling and possess basic language comprehension ability;
5. Ability to understand and willingness to sign informed consent.

Exclusion Criteria:

1. A history of severe diagnosed mental illness (such as depression, anxiety disorder, insomnia);
2. A history of diagnosed cognitive dysfunction (such as intellectual disability, Parkinson's disease);
3. Requires emergency surgery (within 72 hours after diagnosis);
4. Has participated in other interventional clinical trials.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the GAD-7 score (Generalized Anxiety Disorder 7-item Scale) after the Preoperative Communication between Two Groups. | At baseline and 24 hours after routine preoperative communication.
  GAD-7 (Generalized Anxiety Disorder 7-item Scale) is a scale used to assess anxiety-related symptoms. Each of its 7 items is scored from a minimum of 0 to a maximum of 3 points, resulting in a total score ranging from 0 to 21. Higher scores indicate worse outcomes, as they reflect more severe anxiety symptoms.
Change from Baseline in the VAS-A (Visual Analogue Scale-Anxiety) after the Preoperative Communication between Two Groups. | At baseline and 24 hours after routine preoperative communication.
  The VAS-A (Visual Analogue Scale for Anxiety) is a simple scoring tool used to measure the severity of anxiety symptoms. It consists of a single 10-centimeter line with anchors at either end (e.g., "no anxiety" at 0 and "extreme anxiety" at 10). Patients mark a point on the line to indicate their current anxiety level, and the score is measured as the distance from the "no anxiety" end. The minimum score is 0 (indicating no anxiety) and the maximum score is 10 (indicating extreme anxiety). Higher scores mean worse outcomes, as they reflect more severe anxiety symptoms.
Change from Baseline in the MCMQ score (Medical Coping Modes Questionnaire) after the Preoperative Communication between Two Groups | At baseline and 24 hours after routine preoperative communication.
  The MCMQ score (Medical Coping Modes Questionnaire) is a scale designed to assess patients' coping strategies when facing illness. It typically consists of 20 items, with each item scored from 1 (least agreement) to 4 (most agreement), resulting in a total score ranging from 20 (minimum) to 80 (maximum).
  Higher scores alone do not universally indicate better or worse outcomes, as the scale measures three distinct coping dimensions: Confrontation (active engagement), Avoidance (distancing), and Resignation (passive acceptance). Higher scores on "Confrontation" often reflect more adaptive coping (better outcome), while higher scores on "Resignation" may indicate less adaptive coping (worse outcome).
Change from Baseline in the PANAS score (Positive and Negative Affect Schedule) after the Preoperative Communication between Two Groups. | At baseline and 24 hours after routine preoperative communication.
  The Positive and Negative Affect Schedule (PANAS) is a widely used psychological tool to measure an individual's positive and negative emotional states. It consists of 20 items (10 for positive affect, 10 for negative affect), with each item rated on a 5-point scale (1 = "very slightly or not at all" to 5 = "extremely"). For each dimension: the minimum score is 10 (little to no affect) and the maximum score is 50 (intense affect).
  Higher scores on the Positive Affect (PA) subscale indicate better outcomes (e.g., greater enthusiasm, alertness, or joy), while higher scores on the Negative Affect (NA) subscale indicate worse outcomes (e.g., more distress, fear, or anger).

SECONDARY OUTCOMES:
Change from Baseline in the Heart Rate after the Preoperative Communication between Two Groups. | At baseline and 24 hours after routine preoperative communication.
  Heart rate is measured under resting conditions, with two times measured, and the average value is calculated. Heart rate (HR) is defined as the number of heartbeats per minute (bpm), higher HR may signal adverse reactions, or physiological stress.
Change from Baseline in the Blood Pressure after the Preoperative Communication between Two Groups. | At baseline and 24 hours after routine preoperative communication.
  Blood pressure (BP) is recorded as two values: systolic blood pressure (SBP) and diastolic blood pressure (DBP). BP is measured under resting conditions, with two measurements taken, and the average value is calculated. Higher BP value may indicate a more tense state.
Change from Baseline in the PSQ-18 ( Patient Satisfaction Questionnaire-18) after the Preoperative Communication between Two Groups. | At baseline and 24 hours after routine preoperative communication.
  The PSQ-18, or Patient Satisfaction Questionnaire-18, is a scale designed to assess patient satisfaction with healthcare services. It consists of 18 items, each rated on a 5-point Likert scale (1 = "very dissatisfied" to 5 = "very satisfied") to evaluate domains like communication, accessibility, and quality of care.
  The total score ranges from 18 (minimum, indicating very low satisfaction) to 90 (maximum, indicating very high satisfaction).Higher scores on the PSQ-18 mean better outcomes, reflecting greater patient satisfaction with the healthcare experience.
Change from Baseline in the EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) after the Preoperative Communication between Two Groups. | At baseline and 24 hours after routine preoperative communication.
  The EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30) is a widely used self-report scale assessing health-related quality of life (HRQoL) in cancer patients. It comprises 30 items measuring three domains: functional scales (e.g., physical, role, emotional function), symptom scales (e.g., fatigue, pain, nausea), and a global health status/HRQoL scale.
  Scores for each domain are linearly transformed to a range of 0 to 100. For functional scales and the global health status/HRQoL scale, higher scores indicate better outcomes (e.g., better physical function or overall quality of life).
  For symptom scales, higher scores indicate worse outcomes (e.g., more severe fatigue or pain).
Change from Baseline in the APAIS (Amsterdam Preoperative Anxiety and Information Scale) after the Preoperative Communication between Two Groups. | At baseline and 24 hours after routine preoperative communication.
  The APAIS (Amsterdam Preoperative Anxiety and Information Scale) is a tool designed to assess two key aspects of preoperative psychological state: anxiety related to surgery/anesthesia and the need for information about the procedure. It consists of 6 items, with 4 measuring anxiety (e.g., "I am worried about the anesthesia") and 2 assessing information needs (e.g., "I would like more information about what will happen during the operation"). Each item is rated on a 5-point Likert scale (1 = "not at all" to 5 = "extremely").
  The total score ranges from 6 (minimum, indicating very low anxiety and minimal information needs) to 30 (maximum, indicating severe anxiety and strong information needs). Higher scores on the APAIS generally mean worse outcomes, as they reflect greater preoperative anxiety (a negative psychological state) and/or heightened unmet information needs.
Change from Baseline in the B-IPQ-PCa (Brief Illness Perception Questionnaire for Prostate Cancer) after the Preoperative Communication between Two Groups. | At baseline and 24 hours after routine preoperative communication.
  The B-IPQ-PCa (Brief Illness Perception Questionnaire for Prostate Cancer) is a validated tool designed to assess prostate cancer patients' perceptions of their illness. It adapts the original Brief Illness Perception Questionnaire (B-IPQ) to focus on prostate cancer-specific experiences, measuring domains such as perceived illness timeline, consequences, personal/treatment control, identity (symptom burden), concern, emotional impact, and understanding of the illness.
  The scale typically includes 8 scored items rated on 0-10 scale. Total scores range from 0 (minimum, reflecting more positive/adaptive illness perceptions) to 80 (maximum, indicating more negative/maladaptive perceptions).
Difference of the NASA-TLX (NASA Task Load Index) between Two Groups | 1 hour after routine preoperative communication.
  The NASA-TLX (NASA Task Load Index) is a widely used subjective assessment tool designed to measure perceived workload associated with performing a task. It evaluates six dimensions of workload: Mental Demand (cognitive effort), Physical Demand (physical effort), Temporal Demand (time pressure), Performance (self-rated task success), Effort (amount of work invested), and Frustration Level (stress or irritation).
  Each dimension is rated by the participant on a 0-100 scale (0 = "very low" to 100 = "very high"). These ratings are combined to generate an overall workload score, which ranges from 0 (minimum, indicating negligible workload) to 100 (maximum, indicating extreme workload).
  Higher scores on the NASA-TLX mean worse outcomes, as they reflect greater perceived task difficulty, cognitive/physical strain, or stress associated with the task.
Change from Baseline in the GAD-7 score (Generalized Anxiety Disorder 7-item Scale) after the LLM-assisted Preoperative Communication in LLM-assisted Group. | At baseline and 24 hours after LLM-assisted preoperative communication.
  GAD-7 (Generalized Anxiety Disorder 7-item Scale) is a scale used to assess anxiety-related symptoms. Each of its 7 items is scored from a minimum of 0 to a maximum of 3 points, resulting in a total score ranging from 0 to 21. Higher scores indicate worse outcomes, as they reflect more severe anxiety symptoms.
Change from Baseline in the VAS-A (Visual Analogue Scale for Anxiety) Scale after the LLM-assisted Preoperative Communication in LLM-assisted Group. | At baseline and 24 hours after LLM-assisted preoperative communication.
  The VAS-A (Visual Analogue Scale for Anxiety) is a simple scoring tool used to measure the severity of anxiety symptoms. It consists of a single 10-centimeter line with anchors at either end (e.g., "no anxiety" at 0 and "extreme anxiety" at 10). Patients mark a point on the line to indicate their current anxiety level, and the score is measured as the distance from the "no anxiety" end. The minimum score is 0 (indicating no anxiety) and the maximum score is 10 (indicating extreme anxiety). Higher scores mean worse outcomes, as they reflect more severe anxiety symptoms.
Change from Baseline in the MCMQ score (Medical Coping Modes Questionnaire) after the LLM-assisted Preoperative Communication in LLM-assisted Group. | At baseline and 24 hours after LLM-assisted preoperative communication.
  The MCMQ score (Medical Coping Modes Questionnaire) is a scale designed to assess patients' coping strategies when facing illness. It typically consists of 20 items, with each item scored from 1 (least agreement) to 4 (most agreement), resulting in a total score ranging from 20 (minimum) to 80 (maximum). Higher scores alone do not universally indicate better or worse outcomes, as the scale measures three distinct coping dimensions: Confrontation (active engagement), Avoidance (distancing), and Resignation (passive acceptance). Higher scores on "Confrontation" often reflect more adaptive coping (better outcome), while higher scores on "Resignation" may indicate less adaptive coping (worse outcome).
Change from Baseline in the PANAS score (Positive and Negative Affect Schedule) after the LLM-assisted Preoperative Communication in LLM-assisted Group. | At baseline and 24 hours after LLM-assisted preoperative communication.
  The Positive and Negative Affect Schedule (PANAS) is a widely used psychological tool to measure an individual's positive and negative emotional states. It consists of 20 items (10 for positive affect, 10 for negative affect), with each item rated on a 5-point scale (1 = "very slightly or not at all" to 5 = "extremely"). For each dimension: the minimum score is 10 (little to no affect) and the maximum score is 50 (intense affect). Higher scores on the Positive Affect (PA) subscale indicate better outcomes (e.g., greater enthusiasm, alertness, or joy), while higher scores on the Negative Affect (NA) subscale indicate worse outcomes (e.g., more distress, fear, or anger).

CONTACTS AND LOCATIONS:
Overall Officials: Bo Dai, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No